CLINICAL TRIAL: NCT06232408
Title: Phase 1 Trial of the Safety, Pharmacokinetics, Pharmacodynamics, and Preliminary Clinical Activity of RP-1664 in Participants With Advanced Solid Tumors
Brief Title: LIONS (PLK4 Inhibitor in Advanced Solid Tumors)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decided to terminate study early
Sponsor: Repare Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RP-1664-01
Record Dates: First submitted 2024-01-09; First posted 2024-01-30 (Actual); Results first posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- RP-1664 (Experimental)
  Interventions: Drug: RP-1664

INTERVENTIONS:
Drug: RP-1664 — RP-1664 will be supplied as immediate-release solid dosage form for oral self-administration.

SUMMARY:
The primary objective of this study is to identify a safe and tolerated dose and schedule of the orally administered PLK4 inhibitor RP-1664. In addition, this study will examine the pharmacokinetics (PK), pharmacodynamics (PD) and preliminary anti-tumor activity of RP-1664 in advanced solid tumors.

DETAILED DESCRIPTION:
This is a first-in-human, Phase 1, multi-center, open-label, dose-escalation and expansion study to:

Evaluate the safety profile and MTD of RP-1664 and establish a recommended dose and schedule for further clinical investigation, In addition, the study aims to characterize the PK, PD, and preliminary anti-tumor activity of orally administered RP-1664. Exploratory objectives include examination of biomarker responses in relationship to RP-1664 exposure.

After the recommended dose and schedule is determined, expansion cohorts with molecularly selected advanced solid tumors will be enrolled to preliminarily assess the anti-tumor effect, and further examine the safety and PK of RP-1664 at the RP2D.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent or assent, according to local guidelines, signed and dated by the patient or legal guardian prior to the performance of any study-specific procedures, sampling, or analyses.
* Male or female and ≥ 12 years-of-age at the time of signature of the consent or assent, and are at least 6th grade reading level to consent; participants < 18 years of age must weigh at least 40 kg.
* Life expectancy ≥ 4 months.
* Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0 or 1.
* Locally advanced or metastatic solid tumor that has progressed or was nonresponsive or intolerant to available therapies and for which no standard or available curative therapy exists.
* Measurable disease as per RECIST v1.1 or INRC.
* Existing biomarker profile (tumor tissue or plasma) reported from a local test obtained in a CLIA-certified or equivalent laboratory demonstrating eligible tumor biomarkers.
* Available tumor tissue.
* Molecularly eligible tumor profile from a CLIA-certified pathology report.
* Ability to comply with the protocol and study procedures detailed in the Schedule of Assessments.
* Ability to swallow and retain oral medications.
* Acceptable organ function at screening.
* Acceptable blood counts at screening.
* Negative pregnancy test (serum or urine) for females of childbearing potential at Screening and while on study drug.
* Resolution of all toxicities of prior treatment or surgery.
* Use of highly effective forms of contraception.

Exclusion Criteria:

* History or current condition (such as transfusion dependent anemia or thrombocytopenia), therapy, or laboratory abnormality that might confound the study results, or interfere with the patient's participation for the full duration of the study treatment.
* Life-threatening illness, medical condition, active uncontrolled infection, or organ system dysfunction or other reasons which, in the investigator's opinion, could compromise the patient's safety.
* Uncontrolled, symptomatic brain metastases.
* Presence of other known second malignancy with the exception of any cancer that has been in complete remission for ≥ 2 years or completely resected squamous and basal cell carcinomas of the skin.
* Patients with active, uncontrolled bacterial, fungal, or viral infection, including hepatitis B virus (HBV), hepatitis C virus (HCV), known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS) related illness.
* Clinically significant vascular (both arterial and venous) and non-vascular cardiac conditions, active or within 6 months prior to enrollment.
* Moderate or severe hepatic impairment (ie, Child-Pugh class B or C).
* Uncontrolled high blood pressure.
* Chemotherapy, small molecule or biologic antineoplastic agent given within 21 days.
* Previously prescribed receptor activator of nuclear factor kappa B ligand (RANKL) inhibitor initiated less than 4 months prior to trial entry. Bisphosphonates are allowed if initiated/administered at least 28 days prior to enrollment.
* I-131 Meta-Iodo-Benzyl-Guanidine (MIGB) therapy within 6 weeks prior to initiation of trial treatment.
* Prior treatment with a PLK4 inhibitor.
* Current treatment with medications that are known to prolong the QT interval.

Ages: 12 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2024-02-14 (Actual); Primary Completion 2025-08-27 (Actual); Study Completion 2025-08-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (4):
  - Participating Site 1025, San Francisco, California
  - Participating Site 1012, New Haven, Connecticut
  - Participating Site 1008, New York, New York
  - Participating Site 1004, New York, New York
- Participating Site 4001, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vallee F, Casas-Selves M, Bubenik M, Duplessis M, Sow B, Suarez C, Sangiorgi B, Li L, Hyer M, Papp R, Leclaire ME, Perryman AL, Liu B, Surprenant S, Mochirian P, Pau V, Maderova Z, Mader P, Yin SY, Goodfellow E, Roulston A, Stocco R, Godbout C, Baruah P, Bonneau-Fortin A, Schonhoft JD, Nejad P, Norman D, Truong VL, Crane S, Attia MA, Mao D, Sicheri F, Marshall CG, Zimmermann M, Bendahan D, Gallant M, Black WC. Discovery of RP-1664: A First-in-Class Orally Bioavailable, Selective PLK4 Inhibitor. J Med Chem. 2025 Jun 12;68(11):10631-10647. doi: 10.1021/acs.jmedchem.5c00529. Epub 2025 May 16. PMID 40378279

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dose Escalation phase only; Dose expansion was not conducted
Groups:
- 10 mg QD RP-1664, 2w on/1w Off: 10 mg QD oral (PO) RP-1664 daily, on a 2 weeks on and 1 week of schedule (21-day treatment cycle)
- 30 mg QD RP-1664, 2w on/1w Off: 30 mg QD oral (PO) RP-1664 daily, on a 2 weeks on and 1 week of schedule (21-day treatment cycle)
- 40 mg QD RP-1664, 2w on/1w Off: 40 mg QD oral (PO) RP-1664 daily, on a 2 weeks on and 1 week of schedule (21-day treatment cycle)
- 60 mg QD RP-1664, 2w on/1w Off: 60 mg QD oral (PO) RP-1664 daily, on a 2 weeks on and 1 week of schedule (21-day treatment cycle)
- 60 mg QD RP-1664, 1w on/1w Off: 60 mg QD oral (PO) RP-1664 daily, on a 1 week on and 1 week of schedule (28-day treatment cycle)
- 90 mg QD RP-1664, 1w on/1w Off: 90 mg QD oral (PO) RP-1664 daily, on a 1 week on and 1 week of schedule (28-day treatment cycle)
Period: Overall Study
Arm/Group | 10 mg QD RP-1664, 2w on/1w Off | 30 mg QD RP-1664, 2w on/1w Off | 40 mg QD RP-1664, 2w on/1w Off | 60 mg QD RP-1664, 2w on/1w Off | 60 mg QD RP-1664, 1w on/1w Off | 90 mg QD RP-1664, 1w on/1w Off
Started | 1 | 1 | 4 | 3 | 16 | 4
Completed | 1 | 1 | 0 | 1 | 0 | 0
Not Completed | 0 | 0 | 4 | 2 | 16 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 10 mg QD RP-1664, 2w on/1w Off | 30 mg QD RP-1664, 2w on/1w Off | 40 mg QD RP-1664, 2w on/1w Off | 60 mg QD RP-1664, 2w on/1w Off | 60 mg QD RP-1664, 1w on/1w Off | 90 mg QD RP-1664, 1w on/1w Off | Total
Number analyzed (Participants) | 1 | 1 | 4 | 3 | 16 | 4 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 2 | 0 | 2 | 0 | 4
  Between 18 and 65 years | 0 | 1 | 1 | 2 | 9 | 3 | 16
  >=65 years | 1 | 0 | 1 | 1 | 5 | 1 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 84 (0) | 53 (0) | 33.3 (28.34) | 61.7 (14.01) | 45.4 (20.71) | 54.5 (14.20) | 48.3 (21.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 1 | 3 | 12 | 3 | 19
  Male | 1 | 1 | 3 | 0 | 4 | 1 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 1 | 4 | 3 | 16 | 4 | 29
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Treatment Related Treatment-Emergent Adverse Events (TRAE) With ≥3 CTCAE Grade
Description: Number of participants with TRAE
Time Frame: Start of treatment through up to 6 months post last dose (up to 18 months)
Measure: Count of Participants; unit: Participants
Arm/Group | 10 mg QD RP-1664, 2w on/1w Off | 30 mg QD RP-1664, 2w on/1w Off | 40 mg QD RP-1664, 2w on/1w Off | 60 mg QD RP-1664, 2w on/1w Off | 60 mg QD RP-1664, 1w on/1w Off | 90 mg QD RP-1664, 1w on/1w Off
Number analyzed (Participants) | 1 | 1 | 4 | 3 | 16 | 4
Participants | 1 | 0 | 3 | 3 | 9 | 3

2. Primary Outcome: Dose Limiting Toxicities (DLT) to Determine a Maximum Tolerated Dose and Schedule of RP-1664 Based on Safety and Tolerability
Description: The number of participants with DLTs during the DLT observation period
Time Frame: During the first cycle (either 21 or 28 days) following the initiation of the study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | 10 mg QD RP-1664, 2w on/1w Off | 30 mg QD RP-1664, 2w on/1w Off | 40 mg QD RP-1664, 2w on/1w Off | 60 mg QD RP-1664, 2w on/1w Off | 60 mg QD RP-1664, 1w on/1w Off | 90 mg QD RP-1664, 1w on/1w Off
Number analyzed (Participants) | 1 | 1 | 3 | 3 | 13 | 2
Participants | 0 | 0 | 0 | 2 | 0 | 1

ADVERSE EVENTS:
Time Frame: Start of treatment through up to 6 months post last dose (up to 18 months)
Groups:
- 10QD 2/1: 10 mg QD oral (PO) RP-1664 daily, on a 2 weeks on and 1 week of schedule (21-day treatment cycle)
- 30QD 2/1: 30 mg QD oral (PO) RP-1664 daily, on a 2 weeks on and 1 week of schedule (21-day treatment cycle)
- 40QD 2/1: 40 mg QD oral (PO) RP-1664 daily, on a 2 weeks on and 1 week of schedule (21-day treatment cycle)
- 60QD 2/1: 60 mg QD oral (PO) RP-1664 daily, on a 2 weeks on and 1 week of schedule (21-day treatment cycle)
- 60QD 1/1: 60 mg QD oral (PO) RP-1664 daily, on a 1 week on and 1 week of schedule (28-day treatment cycle)
- 90QD 1/1: 90 mg QD oral (PO) RP-1664 daily, on a 1 week on and 1 week of schedule (28-day treatment cycle)
- Total: All patients in study
Arm/Group | 10QD 2/1 | 30QD 2/1 | 40QD 2/1 | 60QD 2/1 | 60QD 1/1 | 90QD 1/1 | Total
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1 | 0/4 | 1/3 | 2/16 | 1/4 | 4/29
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 1/4 | 3/3 | 5/16 | 3/4 | 12/29
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1 | 4/4 | 3/3 | 15/16 | 4/4 | 28/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 10QD 2/1 (N=1) | 30QD 2/1 (N=1) | 40QD 2/1 (N=4) | 60QD 2/1 (N=3) | 60QD 1/1 (N=16) | 90QD 1/1 (N=4) | Total (N=29)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 2
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Device dislocation (Product Issues) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 10QD 2/1 (N=1) | 30QD 2/1 (N=1) | 40QD 2/1 (N=4) | 60QD 2/1 (N=3) | 60QD 1/1 (N=16) | 90QD 1/1 (N=4) | Total (N=29)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 2 | 2 | 6 | 3 | 15
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 3
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 3
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 3 | 2 | 2 | 3 | 11
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 1 | 3 | 1 | 7
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 3 | 1 | 5
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 2
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 2 | 1 | 5
Dental caries (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 2 | 3 | 11 | 3 | 20
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 2 | 1 | 4
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 7 | 2 | 9
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 6 | 1 | 8
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Chills (General disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 2
Fatigue (General disorders) | 1 | 0 | 1 | 1 | 8 | 2 | 13
Localised oedema (General disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 3
Oedema (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 3
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Pyrexia (General disorders) | 0 | 0 | 1 | 1 | 1 | 1 | 4
Abdominal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hordeolum (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Rhinovirus infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 2
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 0 | 0 | 2
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 1 | 1 | 0 | 3
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 2
Weight decreased (Investigations) | 0 | 0 | 1 | 1 | 1 | 1 | 4
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 3 | 2 | 7
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 3
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 1 | 0 | 1 | 1 | 4
Headache (Nervous system disorders) | 0 | 0 | 1 | 1 | 2 | 1 | 5
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Device dislocation (Product Issues) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 7 | 3 | 12
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 3 | 1 | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1 | 3 | 0 | 6
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 6 | 2 | 9
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 2

LIMITATIONS AND CAVEATS:
The study was terminated early.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2025-03-24): https://cdn.clinicaltrials.gov/large-docs/08/NCT06232408/Prot_000.pdf
  • Statistical Analysis Plan (2025-09-10): https://cdn.clinicaltrials.gov/large-docs/08/NCT06232408/SAP_001.pdf